CLINICAL TRIAL: NCT05562895
Title: A Multicenter Study to Evaluate the Cios Spin and the Ion Endoluminal System for Pulmonary Nodule Biopsy
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-ION-002
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects with biopsy of pulmonary nodule using Ion Endoluminal System and Cios Spin: Subjects in which a pulmonary nodule biopsy was attempted or performed with the integrated Ion Endoluminal System and Cios Spin
  Interventions: Device: Ion Endoluminal System and Cios Spin

INTERVENTIONS:
Device: Ion Endoluminal System and Cios Spin — Integrated version of the Ion Endoluminal System and Cios Spin

SUMMARY:
The overall objective of this study is to evaluate procedure characteristics of pulmonary nodule biopsies using the integrated version of Cios Spin and the Ion Endoluminal System.

DETAILED DESCRIPTION:
This study is a post-market, prospective, multicenter, single-arm study of subjects undergoing a pulmonary nodule biopsy using the Ion Endoluminal System in conjunction with the Cios Spin. The aim of the study is to evaluate the integrated version of the two systems. The primary outcomes of the study are focused on evaluating the procedure characteristics of the pulmonary nodule biopsy procedure, including diagnostic yield, sensitivity for malignancy, and rate of tool in nodule.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older at the time of the procedure.
* Pulmonary nodule biopsy attempted/performed using the Ion Endoluminal System and Cios Spin 3D imaging.
* Pulmonary nodule ≤2 cm in largest diameter.
* Subject able to understand and adhere to study requirements and provide informed consent.

Exclusion Criteria:

* Planned lymph node staging performed before nodule biopsy.
* Nodule is a pure ground glass opacity.
* Plan to biopsy multiple nodules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an attempted or performed pulmonary nodule biopsy using the Ion Endoluminal System and Cios Spin, 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Intra-procedure through the 13 month follow up period
  Defined as the sum of true positives and true negatives divided by the total number of nodules (or subjects) biopsied
Sensitivity for malignancy | Intra-procedure through the 13 month follow up period
  Defined as the number of true positives divided by the sum of true positives and false negatives for malignancy
Rate of tool in nodule | Intra-procedure
  Tool in nodule is defined as any portion of the needle visualized within the target in all 3 axes (must be confirmed with 3D imaging)

SECONDARY OUTCOMES:
Total radiation dose | Intra-procedure
  Radiation dose from biopsy procedure, measured by the dose area product (DAP), defined as the product of dose and beam area (Gy cm^2)
Time to achieve tool in nodule | Intra-procedure
  Defined as the time the Ion catheter crosses the endotracheal tube (ETT) to the time tool in nodule is confirmed with 3D imaging

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Casal, MD, Principal Investigator — MD Anderson; Bryan Husta, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, Hillcrest Medical Center, San Diego, California
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - South Austin Hospital, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No